CLINICAL TRIAL: NCT04791020
Title: Topic Cervical Anesthesia Plus Paracervical Blockade vs. Topical Cervical Anesthesia Alone for Pain Control During Endouterine Manual Aspiration
Brief Title: Topic Cervical Anesthesia Plus Paracervical Blockade for Pain Control During Endouterine Manual Aspiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Coordinator of research, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-555
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Pain; Abortion, Spontaneous
Keywords: Endouterine manual aspiration; Paracervical blockade; Lidocaine gel
MeSH Terms: conditions — Pain; Abortion, Spontaneous | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine + paracervical blockade (Active Comparator): 5 minutes previous to endouterine manual aspiration, 5mL of lidocaine gel was applied plus standard paracervical blockade.
  Interventions: Drug: Lidocain topical + paracervical blockade
- Lidocaine (Experimental): 5 minutes previous to endouterine manual aspiration, 5mL of lidocaine gel was applied.
  Interventions: Drug: Lidocaine topical

INTERVENTIONS:
Drug: Lidocain topical + paracervical blockade — 5mL of lidocaine gel applied topically to cervix previous to clamping and paracervical blockade
  Arms: Lidocaine + paracervical blockade
Drug: Lidocaine topical — 5mL of lidocaine gel applied topically to cervix previous to clamping, No paracervical blockade will be applied.
  Arms: Lidocaine

SUMMARY:
To compare the effectiveness of lidocaine gel plus paracervical blockade vs. lidocaine gel alone in the management of pain during endouterine manual aspiration.

ELIGIBILITY:
Inclusion Criteria:

* Need for a endouterine manual aspiration (incomplete abortion or gynecological bleeding).

Exclusion Criteria:

* Allergy to lidocain

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Global evaluation of pain | 5 minutes post procedure
  Visible scale of pain evaluation

SECONDARY OUTCOMES:
Adverse reaction | 5 minutes post procedure
  Presence of adverse effects to the drug used (lidocaine gel)

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Thomas H, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No